CLINICAL TRIAL: NCT03559465
Title: Profibrosing Role of B Lymphocytes in Patients With Systemic Sclerosis.
Acronym: SCLERO-LB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016_63; 2017-A02720-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Scleroderma, Systemic
Keywords: systemic sclerosis; B lymphocyte
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with Scs (Experimental): patients with SSc, (10 diffuse forms and 20 limited forms)
  Interventions: Procedure: skin biopsy; Other: Blood punction
- healthy subject (Sham Comparator)
  Interventions: Other: Blood punction

INTERVENTIONS:
Procedure: skin biopsy — A skin biopsy will be performed in 10 patients in the form of 2 punches of 5 mm in the injured area in aseptic condition with a Rodnan score.
  In this study, 10 skin biopsies are needed, and will be performed on the first 10 patients accepting this biopsy.
  Arms: patient with Scs
Other: Blood punction — 1 blood punction during the normal pathway of care of the patient. This punction will be used to perform the extraction of B lymphocyte

SUMMARY:
B Lymphocytes are thought to play an important role in the pathophysiology of systemic sclerosis. In this study, the profibrosing role of B lymphocytes of patients with systemic sclerosis will be evaluated.

DETAILED DESCRIPTION:
B Lymphocytes of patients with systemic sclerosis will be assessed in term of interaction with fibroblasts from patients with systemic sclerosis and compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

patients

* systemic sclerosis according to ACR-EULAR 2013
* written consent
* available insurance

Healthy "blood" and healthy "biopsy" controls

* written consent
* available insurance

Exclusion Criteria:

patients

* overlap with other connective tissue diseases
* immunosuppressants in the past 12 months
* corticosteroids ≥10mg/d
* pregnancy or breast feeding

Healthy "blood" and healthy "biopsy" controls

* systemic sclerosis according to ACR-EULAR 2013
* another connective tissue diseases
* immunosuppressants in the past 12 months
* corticosteroids ≥10mg/d
* pregnancy or breast feeding
* With dysimmune inflammatory diseases (except thyroiditis)
* Presenting an infection in progress or within the previous 15 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Fibroblast transcriptomic : myofibroblast signature | 36 months
  expression of alpha Smooth Muscle Actin

SECONDARY OUTCOMES:
Fibroblast transcriptomic | 36 months
  expression of COL1A1, COL1A2, COL3A1 by quantitative RT-PCR
Difference in collagen infiltration by PicroSirius red staining between the skin biopsies of the two groups | 36 months
Difference in the inflammatory infiltrate by immunohistological markings between the skin biopsies of the two groups | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France